CLINICAL TRIAL: NCT03402555
Title: Observational Study: Image Collection of Infant/Toddler Stools for Danone Software Development
Brief Title: Study of Stool Patterns to Collect a Panel of Stool Images for the Development of a Software
Acronym: Poobao
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: ObvioHealth (Industry)
Responsible Party: Sponsor
Other Study IDs: EBB17GC16961
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Stool pattern — Collection of stool images

SUMMARY:
Collection of a panel of stool images from healthy infants/toddlers for the development of a software

DETAILED DESCRIPTION:
To collect at least 200 images per Brussels Infant and Toddler Stool Scale (BITSS) score and at least 200 images of empty (no stool) disposable diapers from healthy infants/toddlers aged 0-24 months for the development of a software

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants/toddlers (0-24 months of age at time of enrollment)
2. Informed consent from mother ≥21 years of age
3. In-home access to reliable internet connections; a mobile device suitable for electronic communication; and a device suitable for capturing and transmitting high-quality electronic images as per the PI's discretion
4. Infant/toddler consumes standard, age-appropriate food (breast milk; formula; commercial/homemade baby, table or finger food)
5. Based on the number of stools already acquired per relevant strata at time of enrollment, infant/toddler may or may not be required to regularly produce stools scored as a Score 1, 2, 6 or 7

Exclusion Criteria:

Mothers of Infants/Toddlers:

1. The use of cloth diapers (mothers must commit to using disposable diapers for the duration of the study)
2. Known to have a significant condition (including during pregnancy) that might interfere with the study compliance, as per PI's clinical judgment
3. Deemed likely to be non-compliant with the study protocol, as per PI's clinical judgment

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy subjects aged 0-24 months
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, MD, Principal Investigator — Obvio Health; Seng Hock Quak, MD, Principal Investigator — National University Hospital, Singapore
Locations (2):
- ObvioHealth, Orlando, Florida, United States
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vandenplas Y, Szajewska H, Benninga M, Di Lorenzo C, Dupont C, Faure C, Miqdadi M, Osatakul S, Ribes-Konickx C, Saps M, Shamir R, Staiano A; BITSS Study Group. Development of the Brussels Infant and Toddler Stool Scale ('BITSS'): protocol of the study. BMJ Open. 2017 Mar 29;7(3):e014620. doi: 10.1136/bmjopen-2016-014620. PMID 28360250

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The mother was to complete an eQuestionnaire for eligibility confirmation and upload 3 separate test images of her infant/toddler's stool via ClaimIt within a window of 10 days. The mother and infant/toddler were enrolled if the test images were successfully uploaded and if they met all inclusion criteria and none of the exclusion criteria.
Groups:
- Mother-infant/Toddler Pairs: 96 mother-infant/toddler pairs were enrolled in the study
Period: Overall Study
Arm/Group | Mother-infant/Toddler Pairs
Started | 96
Completed | 91
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: 96 mother-infant/toddler pairs were included in the analysis
Arm/Group | Mother-infant/Toddler Pairs
Number analyzed (Participants) | 96
Age, Continuous [Mean (Full Range); unit: months] — Age for infant, continuous
  months
    Infant/Toddler | 13.3 [0 to 24]
Age, Continuous [Mean (Full Range); unit: years] — Age for mother, continuous
  years | 30.2 [21 to 48]
Sex: Female, Male [Count of Participants; unit: Participants] — For infant/toddler
  Participants
    Female | 50
    Male | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Stool Images Collected
Description: Creation of a database containing at least 1600 pictures of individual diapers:
  * 200 images of diapers with stool per each score (BITSS types 1 to 7)
  * 200 images of empty (no stool) disposable diapers
Time Frame: At least 30 days
Measure: Number; unit: images
Arm/Group | Mother-infant/Toddler Pairs
Number analyzed (Participants) | 96
images | 2731

2. Other Pre Specified Outcome: A Comparison of the Stool Consistency Scores From the Mothers On-study to Re-scores From Mothers (Not Enrolled on Study) Based Only on the Uploaded Images
Description: A comparison of the stool consistency scores from the mothers on-study to re-scores from two mothers (not enrolled on study, Mother #1 and Mother #2) based only on the uploaded images
Time Frame: 30 days
Measure: Number; unit: percentage of agreement
Arm/Group | Mother-infant/Toddler Pairs
Number analyzed (Participants) | 91
percentage of agreement
  Agreement with Mother #1 | 58.0
  Agreement with Mother #2 | 48.5

3. Other Pre Specified Outcome: An Assessment of Mothers' Perceptions of the Usability of the ClaimIt App
Description: An assessment of mothers' perceptions of the usability of the ClaimIt app with ClaimIt Platform Questionnaire
Time Frame: 30 days
Population: 96 pairs enrolled, 91 completed study, 87 completed the study questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Mother-infant/Toddler Pairs
Number analyzed (Participants) | 87
Participants
  Difficult to score stool pictures: No | 78
  Difficult to score stool pictures: Yes | 9

ADVERSE EVENTS:
Time Frame: no timeframe as no AE/SAE is collected
Description: This is an observation study to collect stool images. no invasive procedures are involved. at risk of SAE/AE is not collected
Arm/Group | Mother-infant/Toddler Pairs
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT03402555/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT03402555/SAP_001.pdf
  • Informed Consent Form (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03402555/ICF_002.pdf